CLINICAL TRIAL: NCT02062021
Title: Understanding the Role of Autoimmune Disorders on the Initial Presentation of Cardiovascular Disease: a CALIBER Proposal Using Linked GPRD-MINAP-HES Data
Brief Title: Understanding the Role of Autoimmune Disorders on the Initial Presentation of Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor of Epidemiology and Public Health, University College, London
Other Study IDs: 13_01
Record Dates: First submitted 2014-01-30; First posted 2014-02-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Myocardial Infarction; Ischemic Stroke; Stroke; Subarachnoid Haemorrhage; Venous Thrombosis; Transient Ischemic Attack; Stable Angina Pectoris; Unstable Angina; Heart Failure; Peripheral Arterial Disease; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Myocardial Infarction; Ischemic Stroke; Stroke; Subarachnoid Hemorrhage; Venous Thrombosis; Ischemic Attack, Transient; Angina, Stable; Angina, Unstable; Heart Failure; Peripheral Arterial Disease; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
Autoimmune diseases are diseases in which inappropriate immune responses that have the capability of harming host cells play an important role. Evidence suggests that the presence of certain autoimmune diseases such as rheumatoid arthritis or systematic lupus erythematosus increase the risk of cardiovascular disease (CVD). However, this evidence is inconsistent for autoimmune disorders and no systematic approach has been previously used to study the relationship between a range of common autoimmune disorders and specific forms of cardiovascular diseases such as myocardial infarction, intracerebral and subarachnoid haemorrhage, or venous thrombosis.

The investigators will use linked electronic health records to investigate whether commonly diagnosed autoimmune disorders are associated with increased risk of CVD development and whether effects differ in men and women and change with age.

DETAILED DESCRIPTION:
The linkage of Clinical Practice Research Datalink (CPRD) to the national registry of acute coronary syndromes (the Myocardial Ischaemia National Audit Project, MINAP), Hospital Episode Statistics (HES) and Office for National Statistics (ONS) available through CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records), offers an opportunity to investigate the association between autoimmune disorders and the initial presentation of non-fatal and fatal specific cardiovascular phenotypes. The use of a systematic approach to investigate whether a range of commonly diagnosed autoimmune disorders are independent risk factors for several specific and well defined arterial and venous diseases will help to improve the investigators understanding of the role of autoimmune disorders in development of specific types of CVD in both men and women and in different age groups. It will also provide useful information to improve existing cardiovascular risk prediction methods that are used in clinical practice for patient management.

ELIGIBILITY:
Inclusion Criteria:

* One year prior to study entry
* 18 years or older
* Recorded sex
* Free of symptomatic cardiovascular disease at entry

Exclusion Criteria:

* Prior cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients registered in Clinical Practice Research Datalink (CPRD) practices
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Rate ratios for the associations between presence of autoimmune disorders and initial presentation of myocardial infarction | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Rate ratios for the associations between presence of autoimmune disorders and initial presentation of stroke | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Rate ratios for the associations between presence of autoimmune disorders and initial presentation of stroke and venous thrombosis | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group

SECONDARY OUTCOMES:
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of stable angina | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associations studied:
  overall by sex by age group
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of unstable angina | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of heart failure | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of peripheral arterial disease | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of transient ischemic attack | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group
Hazard ratios for the association between the presence of autoimmune disease and the initial presentation of abdominal aortic aneurysm | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associated studies:
  overall, by sex, by age group

OTHER OUTCOMES:
Cumulative incidence per autoimmune disease status | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 5 years)
  Associations studied:
  overall by sex by age group

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom